CLINICAL TRIAL: NCT00171223
Title: An Extension to a Phase II Study to Determine the Efficacy and Safety of STI571 in Patients With Chronic Myeloid Leukemia Who Are Refractory to or Intolerant of Interferon-Alpha
Brief Title: An Extension Study to Determine the Efficacy and Safety of STI571 in Participants With Chronic Myeloid Leukemia Who Are Refractory to or Intolerant of Interferon-Alpha
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSTI571A0110E2; 2005-001382-33 (EudraCT Number)
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Results first posted 2021-07-22 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Leukemia, Myelogenous, Chronic, BCR-ABL Positive
Keywords: Chronic Myelogenous Leukemia; CML; Philadelphia Chromosome; Accelerated phase; Acute Myelogenous Leukemia; AML; Acute Lymphoblastic Leukemia; ALL; Imatinib mesylate
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Philadelphia Chromosome; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- All Participants With Chronic Myeloid Leukemia (Experimental): Participants received STI571, capsules or tablets, orally, once a day at a dose of 400 mg. During the Core Phase of the study, participants received STI571 daily for up to 12 months. Participants completing 12 months of therapy were eligible to continue treatment in the Extension Phase of the study, and they continued STI571 for as long as the therapy was beneficial or until death, intolerable toxicity or the decision to discontinue by the investigator, whichever came first. (Maximum duration on study was approximately 14 years).
  Interventions: Drug: STI571

INTERVENTIONS:
Drug: STI571 — STI571 oral capsules or tablets.
  Other Names: Imatinib Mesylate

SUMMARY:
During the Core Phase of the study, participants received STI571 at a dose of 400 milligrams (mg) daily for up to 12 months. Participants completing 12 months of therapy were eligible to continue treatment in the Extension Phase of the study provided that, in the opinion of the investigator, they had benefited from treatment with STI571 and there were no safety concerns.

ELIGIBILITY:
Inclusion Criteria:

Participants included in the study were:

* Consenting males or females greater than or equal to (≥)18 years of age with Philadelphia chromosome positive (Ph+) chronic myeloid leukemia (CML).
* With a documented failure of interferon-alpha (IFN) or an IFN-containing therapy, characterized as resistance or refractoriness defined as any of the following:

  * Hematologic Resistance - Failure to achieve a complete hematological response (CHR), lasting for at least 1 month despite 6 or more months of IFN or an IFN-containing regimen, in which IFN was administered at a dose of at least 25 million international units (MIU) per week. During this treatment period the cumulative duration of hydroxyurea therapy may not have exceeded 50% of the treatment period with the IFN-containing regimen.
  * Cytogenetic Resistance - Bone marrow cytogenetics showing ≥65% Ph+ after one year of IFN-based therapy,
  * Cytogenetic Refractoriness - An increase in the Ph+ chromosome in BM cells by at least 30 percentage points (e.g. from 20% to 50%, or from 30% to 60%) confirmed by two samples at least 1 month apart, or an absolute increase to ≥65%,
  * Hematologic Refractoriness - A rising white blood cell count (WBC) [to a level ≥20 x 10^9/L confirmed by two samples taken at least two weeks apart] for participants achieving a complete hematologic response while receiving IFN or an IFN-containing regimen. This regimen must have included IFN at a dose of at least 25 MIU administered per week. During this treatment period the cumulative duration of hydroxyurea therapy may not have exceeded 50% of the treatment period with the IFN-containing regimen.

In this report all refractory populations were referred to as "relapsed" populations.

* With a documented intolerance to IFN therapy defined as a ≥Grade 3 non-hematologic toxicity persisting for at least one month, for participants receiving IFN or an IFN- containing regimen. IFN was to be administered at a dose of at least 25 MIU/week. Participants who were intolerant of IFN were to have been diagnosed ≥6 months prior to the time of entry into the study.

Exclusion Criteria:

Participants excluded from the study were:

* Females of childbearing potential without a negative pregnancy test prior to the initiation of study drug. Barrier contraceptive precautions were to be used throughout the trial in both sexes.
* With serum bilirubin and creatinine concentrations more than twice the upper limit of the normal range (ULN).
* With serum glutamic oxaloacetic transaminase (SGOT) and serum glutamic pyruvic transaminase (SGPT) more than twice the ULN.
* With >15% of blasts or basophils in peripheral blood (PB) or bone marrow (BM).
* With ≥30% of blasts plus promyelocytes in PB or BM.
* With a platelet count of less than (<)100 x 10^9/L.
* With an Eastern Cooperative Oncology Group (ECOG) Performance Status Score ≥3.
* Receiving busulfan within 6 weeks of Day 1.
* Receiving treatment with IFN or cytosine arabinoside (Ara-C) within 14 days of Day 1.
* Receiving treatment with hydroxyurea within 7 days of Day 1.
* Receiving other investigational agents within 28 days of Day 1.
* With prior marrow or stem cell transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 532 (Actual)
Dates: Start 1999-12-06 (Actual); Primary Completion 2013-11-29 (Actual); Study Completion 2013-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (28):
- United States (11):
  - UCLA Medical Center, Los Angeles, California
  - H. Lee Moffet Cancer Center & Research Institute/Univ of South Florida, Tampa, Florida
  - Northwestern Univ meical School/Robert H. Lurie Comprehensive Cancer Center, Chicago, Illinois
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - Dana Faber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Wayne State University/Kamanos Cancer Center, Detroit, Michigan
  - C/O V. Ward - Washington Univ. school of Medicine, St Louis, Missouri
  - New York Presbyterian Hospital, New York, New York
  - Oregon Health & sciences University, Portland, Oregon
  - MD Anderson Cancer Center, University of Texas, Houston, Texas
- France (3):
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Pessac
  - Novartis Investigative Site, Poitiers
- Germany (4):
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Mannheim
- Italy (7):
  - Novartis Investigative Site, Bologna
  - Novartis Investigative Site, Milan
  - Novartis Investigative Site, Monza
  - Novartis Investigative Site, Orbassano
  - Novartis Investigative Site, Pavia
  - Novartis Investigative Site, Rome
  - Novartis Investigative Site, Udine
- Novartis Investigative Site, Basel, Switzerland
- United Kingdom (2):
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Newcastle upon Tyne

RESULTS

PARTICIPANT FLOW:
Groups:
- Hematologic Failure: Participants failed to achieve a complete hematologic response, defined as lasting for at least 1 month despite 6 or more months of an interferon-alpha containing regimen, or had a rising white blood cell count (WBC) [to a level 20 x 10^9/L] confirmed by two samples taken at least two weeks apart after achieving a complete hematological response while receiving an interferon- alpha containing regimen of at least 25 million international units (MIU) per week. Participants received STI571, capsules or tablets, orally, once a day at a dose of 400 milligrams (mg). During the Core Phase of the study, participants received STI571 daily for up to 12 months. Participants completing 12 months of therapy were eligible to continue treatment in the Extension Phase of the study, and they continued STI571 for as long as the therapy was beneficial or until death, intolerable toxicity or the decision to discontinue by the investigator, whichever came first. (Maximum duration on study was approximately 14 years).
- Cytogenetic Failure: Participants' bone marrow (BM) cytogenetics showed greater than or equal to (>=) 65% Philadelphia chromosome positivity after one year of an interferon-alpha containing regimen or an increase in the Philadelphia chromosome positive BM cells by at least 30 percentage points (e.g., from 20% to 50%, or from 30% to 60%) confirmed by two samples at least 1 month apart, or an increase to >= 65%. Participants received STI571, capsules or tablets, orally, once a day at a dose of 400 mg. During the Core Phase of the study, participants received STI571 daily for up to 12 months. Participants completing 12 months of therapy were eligible to continue treatment in the Extension Phase of the study, and they continued STI571 for as long as the therapy was beneficial or until death, intolerable toxicity or the decision to discontinue by the investigator, whichever came first. (Maximum duration on study was approximately 14 years).
- Interferon-alpha Intolerance: Participants demonstrated intolerance to interferon-alpha therapy defined as a documented greater than (>) Grade 3 nonhematologic toxicity persisting for more than 1 month after receiving an interferon-alpha containing regimen of at least 25 MIU/week. Participants must have been more than 6 months from time of diagnosis. Participants received STI571, capsules or tablets, orally, once a day at a dose of 400 mg. During the Core Phase of the study, participants received STI571 daily for up to 12 months. Participants completing 12 months of therapy were eligible to continue treatment in the Extension Phase of the study, and they continued STI571 for as long as the therapy was beneficial or until death, intolerable toxicity or the decision to discontinue by the investigator, whichever came first. (Maximum duration on study was approximately 14 years).
Period: Overall Study
Arm/Group | Hematologic Failure | Cytogenetic Failure | Interferon-alpha Intolerance
Started | 152 | 188 | 192
Completed (Disposition data is reported till end of study.) | 12 | 47 | 22
Not Completed | 140 | 141 | 170
Not completed — Adverse Event (Non-fatal) | 6 | 5 | 19
Not completed — Abnormal Laboratory Value (s) | 4 | 2 | 3
Not completed — Abnormal Procedure | 1 | 0 | 0
Not completed — Unsatisfactory Therapeutic Effect | 57 | 43 | 52
Not completed — No Longer Requires Study Drug (Bone Marrow Transplant) | 2 | 4 | 2
Not completed — Protocol Violation | 2 | 2 | 3
Not completed — Participant Withdrew Consent | 12 | 21 | 15
Not completed — Lost to Follow-up | 5 | 2 | 3
Not completed — Administrative Problems | 4 | 7 | 6
Not completed — Adverse Event (Serious Fatal) | 6 | 8 | 9
Not completed — Not Specified (No Data Collected After Cut-off) | 41 | 47 | 58

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all enrolled participants.
Groups:
- Hematologic Failure: Participants failed to achieve a complete hematologic response, defined as lasting for at least 1 month despite 6 or more months of an interferon-alpha containing regimen, or had a rising WBC (to a level 20 x 10^9/L) confirmed by two samples taken at least two weeks apart after achieving a complete hematological response while receiving an interferon- alpha containing regimen of at least 25 MIU per week. Participants received STI571, capsules or tablets, orally, once a day at a dose of 400 mg. During the Core Phase of the study, participants received STI571 daily for up to 12 months. Participants completing 12 months of therapy were eligible to continue treatment in the Extension Phase of the study, and they continued STI571 for as long as the therapy was beneficial or until death, intolerable toxicity or the decision to discontinue by the investigator, whichever came first. (Maximum duration on study was approximately 14 years).
- Cytogenetic Failure: Participants' BM cytogenetics showed >= 65% Philadelphia chromosome positivity after one year of an interferon-alpha containing regimen or an increase in the Philadelphia chromosome positive BM cells by at least 30 percentage points (e.g., from 20% to 50%, or from 30% to 60%) confirmed by two samples at least 1 month apart, or an increase to >= 65%. Participants received STI571, capsules or tablets, orally, once a day at a dose of 400 mg. During the Core Phase of the study, participants received STI571 daily for up to 12 months. Participants completing 12 months of therapy were eligible to continue treatment in the Extension Phase of the study, and they continued STI571 for as long as the therapy was beneficial or until death, intolerable toxicity or the decision to discontinue by the investigator, whichever came first. (Maximum duration on study was approximately 14 years).
- Interferon-alpha Intolerance: Participants demonstrated intolerance to interferon-alpha therapy defined as a documented > Grade 3 nonhematologic toxicity persisting for more than 1 month after receiving an interferon-alpha containing regimen of at least 25 MIU/week. Participants must have been more than 6 months from time of diagnosis. Participants received STI571, capsules or tablets, orally, once a day at a dose of 400 mg. During the Core Phase of the study, participants received STI571 daily for up to 12 months. Participants completing 12 months of therapy were eligible to continue treatment in the Extension Phase of the study, and they continued STI571 for as long as the therapy was beneficial or until death, intolerable toxicity or the decision to discontinue by the investigator, whichever came first. (Maximum duration on study was approximately 14 years).
- Total: Total of all reporting groups
Arm/Group | Hematologic Failure | Cytogenetic Failure | Interferon-alpha Intolerance | Total
Number analyzed (Participants) | 152 | 188 | 192 | 532
Age, Continuous [Median (Full Range); unit: years] | 55.5 [18 to 79] | 53.0 [23 to 77] | 59.0 [20 to 90] | 57.0 [18 to 90]
Age, Customized [Count of Participants; unit: Participants]
  Less than (<) 50 years | 57 | 64 | 47 | 168
  >= 50 to <= 60 years | 38 | 65 | 50 | 153
  >= 60 to <= 70 years | 47 | 44 | 68 | 159
  >= 70 years | 10 | 15 | 27 | 52
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 77 | 94 | 221
  Male | 102 | 111 | 98 | 311

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Cytogenetic Response (Complete Cytogenetic Response and Major Cytogenetic Response) to STI571
Description: Response was evaluated from bone marrow aspirates and biopsy samples. Bone marrow cytogenetic studies were performed every 3 months during the core phase of the study, then twice yearly, then annually to evaluate Philadelphia chromosome positive (Ph+). Cytogenetic response was defined as the best response the participant achieved during study. Based on the percentage of Ph+ cells = (positive cells/ examined cells) x100, at each BM assessment the cytogenetic response was classified as: Complete Cytogenetic Response (CCyR):, 0% Ph+ cells; Partial Cytogenetic Response (PCyR):, >0 - 35% Ph+ cells; Minor: >35 - 65% Ph+ cells; and Minimal: >65 - 95% Ph+ cells, None: >95 % Ph+ cells and Not done: <20 metaphases were examined and/or response could not be assigned. Major Cytogenetic Response (MCyR) was defined as sum of the CCyR plus PCyR rates.
Time Frame: Up to 6 years after the start of treatment
Population: Intent-To-Treat (ITT) population included all enrolled participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Hematologic Failure | Cytogenetic Failure | Interferon-alpha Intolerance
Number analyzed (Participants) | 152 | 188 | 192
percentage of participants
  Complete Cytogenetic Response | 29.6 [22.5 to 37.5] | 37.2 [30.3 to 44.6] | 45.8 [38.6 to 53.2]
  Major Cytogenetic Response | 45.4 [37.3 to 53.7] | 63.8 [56.5 to 70.7] | 65.6 [58.4 to 72.3]

2. Secondary Outcome: Percentage of Participants With Complete Hematologic Response to STI571
Description: Hematologic response was evaluated from hematology measurements in the peripheral blood. Complete hematological response was defined as normalization of peripheral blood counts [WBC and platelet count < upper limit of normal (ULN) at the laboratory where the analysis was performed], with a normal WBC differential, and no immature granulocytes present, lasting for 4 weeks.
Time Frame: 12 months after the start of treatment
Population: ITT population included all enrolled participants. Here, overall number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Hematologic Failure | Cytogenetic Failure | Interferon-alpha Intolerance
Number analyzed (Participants) | 143 | 184 | 176
percentage of participants | 94.1 [89.1 to 97.3] | 97.9 [94.6 to 99.4] | 91.7 [86.8 to 95.2]

3. Secondary Outcome: Duration of Complete Hematologic Response to STI571
Description: Duration of hematologic response was defined as the time from the first documentation of the complete hematologic response to the date the loss of complete hematologic response is documented. Loss of complete hematological response was defined as a rising WBC count (increased to a level above the ULN at the laboratory where the analysis was performed confirmed by two samples obtained one month apart). The mean survival time and its standard error were underestimated because the largest observation was censored and the estimation was restricted to the largest event time. Complete hematological response was defined as normalization of peripheral blood counts (WBC and platelet count < ULN at the laboratory where the analysis was performed), with a normal WBC differential, and no immature granulocytes present, lasting for 4 weeks.
Time Frame: 12 months after the start of treatment
Population: as for outcome 2
Measure: Mean (Standard Error); unit: months
Arm/Group | Hematologic Failure | Cytogenetic Failure | Interferon-alpha Intolerance
Number analyzed (Participants) | 143 | 184 | 176
months | 19.3672 (0.6383) | 23.9389 (0.506) | 24.6818 (0.6507)

4. Secondary Outcome: Time to Complete Hematologic Response to STI571
Description: Time to Complete Hematologic Response was defined for all participants with calculated confirmed complete hematologic response as the time until first documented response (which was confirmed >= 4 weeks). Complete hematological response was defined as normalization of peripheral blood counts (WBC and platelet count < ULN at the laboratory where the analysis was performed), with a normal WBC differential, and no immature granulocytes present, lasting for 4 weeks.
Time Frame: 12 months after the start of treatment
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Hematologic Failure | Cytogenetic Failure | Interferon-alpha Intolerance
Number analyzed (Participants) | 143 | 184 | 176
months | 1.64 [0.6 to 2.8] | 0.72 [0.3 to 2.8] | 0.72 [0.3 to 2.8]

5. Secondary Outcome: Number of Participants With Common Toxicity Criteria Grade 3 or 4 Cancer-related Symptoms
Description: National Cancer Institute (NCI)/ National Institute of Health (NIH) provides a grading (severity) scale for each adverse event (AE) term, the Common Toxicity Criteria (CTC). Grade 3 refers to severe AE and Grade 4 refers to life-threatening or disabling AE. Cancer-related symptoms included fever, night sweats, bone pain, arthralgia, abdominal discomfort, fatigue and anorexia.
Time Frame: Up to 9 months after the start of treatment
Population: ITT population included all enrolled participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Hematologic Failure | Cytogenetic Failure | Interferon-alpha Intolerance
Number analyzed (Participants) | 152 | 188 | 192
Participants
  Abdominal Discomfort Grade 3 | 0 | 0 | 0
  Abdominal Discomfort Grade 4 | 0 | 0 | 0
  Anorexia Grade 3 | 0 | 0 | 0
  Anorexia Grade 4 | 0 | 0 | 0
  Arthralgia Grade 3 | 0 | 0 | 1
  Arthralgia Grade 4 | 0 | 0 | 0
  Bone Pain Grade 3 | 0 | 1 | 0
  Bone Pain Grade 4 | 0 | 0 | 0
  Fatigue Grade 3 | 1 | 0 | 0
  Fatigue Grade 4 | 0 | 0 | 0
  Fever Grade 3 | 0 | 0 | 0
  Fever Grade 4 | 0 | 0 | 0
  Night Sweats Grade 3 | 0 | 0 | 0
  Night Sweats Grade 4 | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With Grade 3 or 4 Eastern Cooperative Oncology Group (ECOG) Performance Status
Description: The ECOG performance status was recorded at baseline and every 3 months during the core study. The ECOG Performance Scale has 5 grades. 0 = Fully active, able to carry out all pre-disease activities; 1 = Restricted in strenuous activity but ambulatory and able to carry out work of light or sedentary nature; 2 = Ambulatory and capable of all self-care but unable to carry out work activities. Active about 50% of waking hours; 3 = Capable of limited self-care, confined to bed/chair more than 50% of waking hours; 4 = Completely disabled; cannot carry on self-care. Totally confined to bed/chair.
Time Frame: Up to 9 months after the start of treatment
Population: ITT population included all enrolled participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Hematologic Failure | Cytogenetic Failure | Interferon-alpha Intolerance
Number analyzed (Participants) | 152 | 188 | 192
Participants
  Grade 3 | 1 | 0 | 0
  Grade 4 | 0 | 0 | 0

7. Secondary Outcome: Percentage of Participants Alive Over Time Based on Kaplan-Meier Estimates
Description: Overall survival was defined as the time from the first dose of STI571 to the death of the participant. If a participant is not known to have died, survival was censored at the time of last contact. Kaplan-Meier estimates of the percentage of participants at each time point was calculated.
Time Frame: 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144 and 156 months
Population: ITT population included all enrolled participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Hematologic Failure | Cytogenetic Failure | Interferon-alpha Intolerance
Number analyzed (Participants) | 152 | 188 | 192
percentage of participants
  12 Months | 94.7 [89.8 to 97.3] | 98.9 [95.8 to 99.7] | 97.4 [93.9 to 98.9]
  24 Months | 88.1 [81.8 to 92.3] | 93.6 [89 to 96.3] | 89.5 [84.3 to 93.1]
  36 Months | 84 [77.1 to 89] | 91.5 [86.5 to 94.7] | 83.8 [77.7 to 88.3]
  48 Months | 78.4 [70.9 to 84.2] | 87.1 [81.4 to 91.2] | 76.3 [69.6 to 81.7]
  60 Months | 73.3 [65.2 to 79.7] | 83.8 [77.6 to 88.4] | 73.6 [66.7 to 79.3]
  72 Months | 70.1 [61.9 to 76.9] | 79.7 [73.1 to 84.9] | 71.4 [64.3 to 77.3]
  84 Months | 68.5 [60 to 75.5] | 79.7 [73.1 to 84.9] | 67.2 [59.9 to 73.5]
  96 Months | 66.5 [57.9 to 73.8] | 79.1 [72.3 to 84.3] | 65.9 [58.6 to 72.3]
  108 Months | 63.3 [54.3 to 71] | 78.4 [71.6 to 83.7] | 65.3 [57.9 to 71.7]
  120 Months | 61 [51.8 to 69] | 77 [70 to 82.5] | 63.8 [56.3 to 70.4]
  132 Months | 59.7 [50.4 to 67.9] | 75.4 [68.2 to 81.2] | 62.3 [54.6 to 69]
  144 Months | 57 [47.2 to 65.5] | 73.8 [66.4 to 79.8] | 60.8 [53 to 67.6]
  156 Months | 55.5 [45.6 to 64.3] | 70.1 [62.1 to 76.7] | 60.8 [53 to 67.6]

ADVERSE EVENTS:
Time Frame: Up to approximately 14 years
Description: Safety population included all participants who received at least 1 dose of study drug. Serious adverse events were not collected separately for each disease group (hematologic failure, cytogenetic failure and interferon-alpha intolerant) of participants. All the participants were properly combined for analysis, regardless of the disease groups. Other non-serious adverse events were not collected during the extension phase within the clinical database.
Arm/Group | All Participants With Chronic Myeloid Leukemia
Serious Adverse Events (participants affected / at risk) | 13/532
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants With Chronic Myeloid Leukemia (N=532)
Hip fracture (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Head injury (Injury, poisoning and procedural complications) | 1
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Atrial fibrillation (Cardiac disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Generalised oedema (General disorders) | 1
Anal fistula (Gastrointestinal disorders) | 1
Inflammatory bowel disease (Gastrointestinal disorders) | 1
Gastrointestinal pain (Gastrointestinal disorders) | 1
Mental disorder (Psychiatric disorders) | 1
Pollakiuria (Renal and urinary disorders) | 1
Sepsis (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.